CLINICAL TRIAL: NCT04691427
Title: Effectiveness of Vision Therapy in a Virtual Reality Headset
Brief Title: Effectiveness of Virtual Reality Vision Therapy - VERVE
Acronym: VRVT - VERVE
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: OculoMotor Technologies (Industry)
Collaborators: New Jersey Institute of Technology (Other); Salus University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OMT-01
Record Dates: First submitted 2020-12-15; First posted 2020-12-31 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Convergence Insufficiency
MeSH Terms: conditions — Ocular Motility Disorders

STUDY DESIGN:
Masking Description: Examiner (Outcomes Assessor) will be masked by pooling participants from another study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Active Virtual Reality-Based Vision Therapy (Experimental): Virtual reality vision therapy where participants will be playing a custom-designed video game to act as a therapeutic intervention on a consumer-available virtual reality headset.
  Interventions: Device: Virtual Eye Rotation Vision Exercises (VERVE)

INTERVENTIONS:
Device: Virtual Eye Rotation Vision Exercises (VERVE) — A video game designed with elements of vision therapy will be delivered to participants utilizing consumer-available virtual reality headsets (VIVE Pro Eye).

SUMMARY:
The purpose of this research study is to see how well the treatment of a participant's eye coordination and/or focusing problems improves eye muscle responses and symptoms of eyestrain. We will use an entertainment device called a virtual reality headset to play a custom-designed video game to find out how well the treatment of binocular vision improves a participant's coordination and/or focusing problem. The virtual reality headset uses eye-trackers to monitor progress in a totally objective manner. Objective testing allows the doctor to determine the results without relying on a participant's ability to answer questions or respond verbally in any way. We will compare the results of a participant before and after playing the video game.

ELIGIBILITY:
Inclusion Criteria:

* Age 9 years and older
* CISS score ≥ 16
* Best-corrected distance visual acuity of 20/25 or better in each eye
* Random dot stereopsis appreciation of 500 seconds of arc or better
* Parent or subject understands the protocol and is willing to enroll in the study

Exclusion Criteria:

* Constant strabismus at distance or near
* Vertical heterophoria ≥ 2 ∆ at distance or near
* ≥ 2 line interocular difference in best-corrected visual acuity
* Near point of accommodation > 20 cm in either eye as measured by push-up method
* Manifest or latent nystagmus
* Non-strabismic binocular vision and accommodative disorders associated with known disease of the brain
* Diseases known to affect accommodation, vergence, or ocular motility such as multiple sclerosis, Graves orbitopathy, myasthenia gravis, diabetes mellitus, Parkinson disease
* Any ocular or systemic medication known to affect accommodation or vergence such as anti-anxiety agents (e.g., Librium or Valium), anti-arrhythmic agents (e.g., Cifenline, Cibenzoline), anti-cholinergics, bladder spasmolytic drugs (e.g., Propiverine), hydroxychloroquine, chloroquine, phenothiazines (e.g., Compazine, Mellaril, Thorazine), tricyclic antidepressants (e.g., Elavil, Nortriptyline, Tofranil)
* Inability to comprehend and/or perform any study-related test or procedure

Ages: 9 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-10-14 (Actual); Primary Completion 2024-08-28 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Positive Fusional Vergence | up to 4 weeks post-therapy
  Normal range is >15 Prism Diopters
Near Point of Convergence | up to 4 weeks post-therapy
  Normal range is < 6 cm

SECONDARY OUTCOMES:
Convergence Insufficiency Symptom Survey (CISS) | up to 4 weeks post-therapy
  Normal range is < 21 for adults and < 16 for pediatrics
Vision Quality of Life with Time Survey (VisQuaL-T) | up to 4 weeks post-therapy
  Normal range is > 2.5
Core Elements of Gaming Experience Questionnaire | up to 4 weeks post-therapy
  User experience rating

CONTACTS AND LOCATIONS:
Overall Officials: Chang Yaramothu, PhD, Study Chair — OculoMotor Technologies; Tara L Alvarez, PhD, Principal Investigator — OculoMotor Technologies; Mitchell M Scheiman, OD, PhD, Principal Investigator — OculoMotor Technologies
Locations (2):
- United States (2):
  - OculoMotor Technologies, Newark, New Jersey
  - The Eye Institute at Salus University, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No